CLINICAL TRIAL: NCT05752656
Title: Short- and Long-term Behavioral, Cognitive and Motor Outcomes of Frameless Deep Brain Stimulation in Patients With Parkinson's Disease: a Prospective Observational Study
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4578
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Clinical examinations — Clinical examinations and administration of clinical scales

SUMMARY:
The main objective of the study is to evaluate the improvement in quality of life after deep brain stimulation surgery with frameless technique by comparing the PDQ-39 scale score at baseline (before surgery) and one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic Parkinson's disease according to Movement Disorder Society (MDS) criteria;
* patients who are candidates for deep brain stimulation intervention, according to the international criteria of the "Core assessment program for surgical interventional therapies in Parkinson's disease" (CAPSIT-PD).

Exclusion Criteria:

- patients unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by Parkinson's disease and candidates to intervention of deep brain stimulation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2034-01-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of quality of life | One year
  Evaluation of the PDQ-39 scale score at baseline (before surgery) and one year after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Flavia Torlizzi, Rome, Italy